CLINICAL TRIAL: NCT07366697
Title: Beyond Observation: Validating the Ecological Relevance of the Ad-AHA Stroke Using Sensor-Based Measures
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Professor of Rehabilitation Sciences, KU Leuven
Other Study IDs: s70965
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Upper Limb Motor Impairment; Bimanual Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sensor-based monitoring and clinical assessment — Participants will complete the Ad-AHA Stroke assessment and wear bilateral wrist accelerometers for 3 days to measure real-life bimanual activity. No treatment or experimental intervention will be administered.

SUMMARY:
After a stroke, many people experience difficulty using both hands together in daily life. Most rehabilitation assessments, however, only measure how the affected arm performs in one-handed tasks. This makes it difficult to understand how well people actually use their hands in real-world activities, which are usually bimanual.

The Adult Assisting Hand Assessment - Stroke version (Ad-AHA Stroke) is a new clinical test that evaluates how the affected hand performs during two-handed tasks. While promising, it is still unknown whether the score on this test truly reflects how stroke survivors use their hands in daily life.

This study aims to investigate this question by comparing Ad-AHA Stroke scores with real-life data on hand use, recorded over three days using wrist-worn sensors on both arms. By combining clinical and sensor-based measures, this study will help determine whether the Ad-AHA Stroke can accurately represent everyday bimanual performance after stroke.

DETAILED DESCRIPTION:
This is a single-center, cross-sectional observational study designed to examine the relationship between Ad-AHA Stroke scores and real-life bimanual hand use derived from accelerometry data in chronic stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study procedures.
* Age between 18 and 80 years (inclusive).
* Unilateral supratentorial stroke involving cortical or subcortical structures.
* At least 6 months post-stroke at the time of inclusion.
* Community-dwelling (discharged from hospital and currently living at home).
* Able and willing to wear bilateral wrist-worn sensors (triaxial accelerometers) for three consecutive days.
* Presence of clinically observable bimanual impairment.

Exclusion Criteria:

* Severe upper limb impairment, defined as a Fugl-Meyer Assessment of Upper Extremity (FMA-UE) score ≤ 15.
* Severe cognitive or language comprehension impairment interfering with understanding of study instructions or task performance, as judged during screening.
* Presence of other neurological or orthopedic conditions affecting upper limb function (e.g., Parkinson's disease, multiple sclerosis, severe osteoarthritis, brachial plexus injury).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be adults with chronic stroke (≥ 6 months post-onset) who have observable difficulties in performing bimanual tasks. Participants will be recruited from KU Leuven's rehabilitation network, including university-affiliated rehabilitation centers and outpatient clinics in the Leuven region. All participants will be community-dwelling and medically stable at the time of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between Ad-AHA Stroke total score and accelerometer-derived Use Ratio | Baseline (measurement visit), including a continuous 72-hour wrist accelerometer monitoring period
  The primary endpoint is the strength of association between the Ad-AHA Stroke total score, obtained during the measurement visit, and real-world bimanual upper limb use, quantified by the accelerometer-derived Use Ratio calculated from the subsequent 3-day home monitoring period. The Use Ratio is calculated as the total duration of activity of the affected limb divided by that of the non-affected limb (range 0-1, with 1 indicating equal use of both limbs). This measure reflects spontaneous bimanual activity balance and serves as the primary indicator of the ecological validity of the Ad-AHA Stroke.

SECONDARY OUTCOMES:
Correlation between Ad-AHA Stroke score and composite accelerometer index | Baseline (measurement visit), including a continuous 72-hour wrist accelerometer monitoring period
  The secondary endpoint is the correlation between Ad-AHA Stroke scores and a composite accelerometer index derived from multiple sensor-based features (e.g., Use Ratio, Activity Symmetry Index, Bimanual Bouts, Percentage of Bimanual Time, Median Bilateral Magnitude, Median Magnitude Ratio). The composite index will be constructed using feature selection techniques (e.g., principal component analysis or correlation-based filtering). Spearman's ρ will be used to examine the strength of the association.

OTHER OUTCOMES:
Correlations between Ad-AHA Stroke score and individual accelerometry-derived features | Baseline (measurement visit), including a continuous 72-hour wrist accelerometer monitoring period
  Exploratory analyses will examine the associations between Ad-AHA Stroke total scores and individual accelerometer-derived features, including Activity Symmetry Index (ASI), Number of Bimanual Bouts, Percentage of Bimanual Time, Median Bilateral Magnitude, and Median Magnitude Ratio (MMR). Each metric captures a different dimension of bimanual use symmetry and intensity. Associations will be analyzed using Pearson's r or Spearman's ρ, depending on data distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Principal Investigator — KU Leuven
Locations (1):
- Department of Rehabilitation Sciences, KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided